CLINICAL TRIAL: NCT03744845
Title: The Use of Virtual Reality to Reduce Anxiety and Pain in Perioperative Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-22021
Record Dates: First submitted 2018-05-24; First posted 2018-11-16 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Perioperative Pain; Perioperative Anxiety
Keywords: Pain; Anxiety; Intraoperative Care
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Usual anesthetic care.
- Virtual Reality Intervention Group (Experimental): Virtual Reality Distraction
  Interventions: Other: Virtual Reality Distraction

INTERVENTIONS:
Other: Virtual Reality Distraction — This RCT will utilize an Oculus Go VR headset that delivers VR images and sound. Users will wear the VR headset. A research coordinator will familiarize patients with hardware before use. The VR will be used preoperatively and intraoperatively to distracts patients, and aid with the treatment of pain and anxiety.
  Arms: Virtual Reality Intervention Group

SUMMARY:
We will investigate whether the use of Virtual Reality (VR) preoperatively and intraoperatively can help treat pain and anxiety, as measured by patient feedback, vital signs trends, and the amounts of anesthetics, pain medications and anxiolytics used during surgical procedures. The VR intervention will be studied during short hand surgeries normally performed using local anesthesia and sedation.

DETAILED DESCRIPTION:
Virtual Reality (VR) is a powerful and inexpensive technology that has been effectively used in healthcare settings to treat anxiety and pain, with minimal side effects. In the last two decades, opioid abuse and deaths related to opioids have increased, and opioid naive patients are at increased risk of opioid abuse when opioids are used during their surgical procedures. In addition, anesthetics, anxiolytics and analgesics, namely opioids, have a myriad of side effects that worsen patient experience, and lead to complications and increased costs. There are limited studies on the use of VR in the perioperative setting. Our study is a randomized controlled trial to investigate the use of VR to treat anxiety and pain in perioperative settings. We will recruit 56 patients, 28 in the control group and 28 in the VR group, undergoing short (<2 hrs) hand or upper extremity surgeries under local anesthesia and monitored anesthesia care (MAC). The control group will receive standard anesthetic management and the VR group will be exposed to VR in the preoperative setting and during the surgical procedure, using the clinically validated AppliedVR software. The data collected will included satisfaction questionnaires and pain scores for anxiety/pain pre- and post- procedure, vital signs trends to assess sympathetic response during surgery, and amount of anesthetics used. We hypothesize that the VR group will show decreased anxiety and pain, increased satisfaction, and decreased use of anesthetics during the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older and less or equal to 75 years old.
2. ASA physical status I-II.
3. English speaking.
4. Undergoing elective surgery with local anesthetic with sedation.
5. Surgical time less than 2 hours.

Exclusion Criteria:

1. ASA physical status III or above.
2. Allergy to fentanyl, midazolam or propofol.
3. History of seizure, migraines.
4. Chronic Pain Syndrome.
5. Use of high dose opioids or long acting opioids.
6. Severe anxiety, on daily anxiolytics.
7. Psychiatric comorbidities that preclude the use of VR.
8. Physical disabilities that preclude the use of VR technology in a comfortable manner.
9. Patient refusal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Pre-Op Numeric Rating Scale for Pain | 1 minute during pre-op period
  Self-reported pain intensity pre- and post-operation. Each item is scored 0-10 (0 = no pain, 10 = pain as bad as it can be).
Pre-Op Numeric Rating Scale for Anxiety | 1 minute during pre-op period
  Self-reported anxiety intensity pre-operation. Each item is scored 0-10 (0 = no anxiety, 10 = anxiety as bad as it can be).
Post-Op Numeric Rating Scale for Pain | 1 minute during PACU stay
  Self-reported pain intensity post-operation. Each item is scored 0-10 (0 = no pain, 10 = pain as bad as it can be).
Post-Op Numeric Rating Scale for Anxiety | 1 minute during PACU stay
  Self-reported anxiety intensity post-operation. Each item is scored 0-10 (0 = no anxiety, 10 = anxiety as bad as it can be).
Preoperative Medication Dosage | up to 2 hours during pre-op period
  The amount of midazolam (milligrams [mg]), opioids (mg or micrograms [mcg]), propofol (mg), and other sedatives administered to the patient prior to surgery.
Intraoperative Medication Dosage | up to 2 hours during surgery
  The amount of midazolam (milligrams [mg]), opioid (mg or micrograms [mcg]), propofol (mg), and other sedatives (mg) administered to the patient during surgery.
Postoperative Medication Dosage | approximately 1 hour during PACU stay
  The amount of midazolam (milligrams [mg]), opioid (mg or micrograms [mcg]), propofol (mg), and other sedatives (mg) administered to the patient after surgery.

SECONDARY OUTCOMES:
Blood Pressure | up to 2 hours during surgery
  Systolic and diastolic blood pressure (mmHg)
Heart Rate | up to 2 hours during surgery
  Beats per minute (bpm)
Satisfaction with Anesthesia Survey | 5 minutes during PACU stay
  An instrument that measures patient satisfaction with anesthesia care through open-ended and ranked response questions.
Virtual Reality (VR) Survey | 5 minutes during PACU stay
  An instrument designed by study staff to collect information on patients' experience wearing the VR device. The 16-question survey utilizes free-responses, yes/no, and ranked responses.

CONTACTS AND LOCATIONS:
Overall Officials: Sakura Kinjo, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Orthopedic Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maples-Keller JL, Bunnell BE, Kim SJ, Rothbaum BO. The Use of Virtual Reality Technology in the Treatment of Anxiety and Other Psychiatric Disorders. Harv Rev Psychiatry. 2017 May/Jun;25(3):103-113. doi: 10.1097/HRP.0000000000000138. PMID 28475502
- [Background] Mott J, Bucolo S, Cuttle L, Mill J, Hilder M, Miller K, Kimble RM. The efficacy of an augmented virtual reality system to alleviate pain in children undergoing burns dressing changes: a randomised controlled trial. Burns. 2008 Sep;34(6):803-8. doi: 10.1016/j.burns.2007.10.010. Epub 2008 Mar 5. PMID 18325675
- [Background] Furman E, Jasinevicius TR, Bissada NF, Victoroff KZ, Skillicorn R, Buchner M. Virtual reality distraction for pain control during periodontal scaling and root planing procedures. J Am Dent Assoc. 2009 Dec;140(12):1508-16. doi: 10.14219/jada.archive.2009.0102. PMID 19955069
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Mavridou P, Dimitriou V, Manataki A, Arnaoutoglou E, Papadopoulos G. Patient's anxiety and fear of anesthesia: effect of gender, age, education, and previous experience of anesthesia. A survey of 400 patients. J Anesth. 2013 Feb;27(1):104-8. doi: 10.1007/s00540-012-1460-0. Epub 2012 Aug 3. PMID 22864564
- [Background] Soelberg CD, Brown RE Jr, Du Vivier D, Meyer JE, Ramachandran BK. The US Opioid Crisis: Current Federal and State Legal Issues. Anesth Analg. 2017 Nov;125(5):1675-1681. doi: 10.1213/ANE.0000000000002403. PMID 29049113
- [Background] West NA, Severtson SG, Green JL, Dart RC. Trends in abuse and misuse of prescription opioids among older adults. Drug Alcohol Depend. 2015 Apr 1;149:117-21. doi: 10.1016/j.drugalcdep.2015.01.027. Epub 2015 Jan 31. PMID 25678441
- [Background] Sun EC, Darnall BD, Baker LC, Mackey S. Incidence of and Risk Factors for Chronic Opioid Use Among Opioid-Naive Patients in the Postoperative Period. JAMA Intern Med. 2016 Sep 1;176(9):1286-93. doi: 10.1001/jamainternmed.2016.3298. PMID 27400458
- [Background] Chan PY, Scharf S. Virtual Reality as an Adjunctive Nonpharmacological Sedative During Orthopedic Surgery Under Regional Anesthesia: A Pilot and Feasibility Study. Anesth Analg. 2017 Oct;125(4):1200-1202. doi: 10.1213/ANE.0000000000002169. PMID 28598921
- [Background] Pandya PG, Kim TE, Howard SK, Stary E, Leng JC, Hunter OO, Mariano ER. Virtual reality distraction decreases routine intravenous sedation and procedure-related pain during preoperative adductor canal catheter insertion: a retrospective study. Korean J Anesthesiol. 2017 Aug;70(4):439-445. doi: 10.4097/kjae.2017.70.4.439. Epub 2017 Mar 15. PMID 28794840